CLINICAL TRIAL: NCT06200090
Title: Empathy and Emotional Regulation as Protective Factors Against Burnout Among Nursing Students: A Multi-National Cross-Sectional Study
Brief Title: Empathy and Emotional Regulation: A Multi-National Cross-Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Associate Professor, Mansoura University
Other Study IDs: EmpathyMulti-National7
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Empathy; Emotional Regulation; Burnout
MeSH Terms: conditions — Emotional Regulation; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Significant levels of psychological disorders and psychological distress among higher education students have been reported worldwide (Galdino et al., 2020), given that during these years there is a peak in prevalence of many mental disorders, particularly major depressive disorder (18.5% to 21.2%), generalized anxiety disorder (18.6% to 16.7%) and drug use disorder (45.9% to 59.8%). (Auerbach et al., 2018). Additionally, compared to other major students, medical school and nursing students experienced higher levels of burnout due to the complex curriculum and pressure for professional performance (Ling et al., 2014). Altogether, this evidence show that nursing students frequently experience psychological and emotional problems such as academic exhaustion, stress, depression, and anxiety during their four years of completing their degree (Hwang & Kim, 2022).

To the best of our knowledge, this study is the first of its kind that addresses the issue of burnout and its relation to empathy and emotional regulation among nursing students at the middle east. Analyzing burnout syndrome among undergraduate nursing students may provide support for managers to implement prevention and management strategies in relation to the syndrome, in order to ensure health and well-being during the professional training process, as well as providing training for nurses engaged and prepared to provide quality care. Thus, this study aims to investigate the burnout syndrome among nursing students and its relation to empathy and emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students from the five full-time levels

Exclusion Criteria:

-

Ages: 17 Years to 27 Years | Sex: All
Age Groups: Child, Adult
Study Population: Undergraduate nursing students from the five full-time levels
Sampling Method: Non-Probability Sample
Enrollment: 1987 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Inventory-Student Survey (MBI-SS) | Baseline
  The MBI-SS is made up of 15 items that constitute three scales: emotional exhaustion (EX; five items), cynicism (CY; four items), and academic efficacy (AE; six items). All the items are scored by using a seven-point Likert scale [from 0 (never) to 6 (always)]. High scores on EX, CY and low scores on AE were indicative of burnout (Academic efficacy items are reversed scored). According to the MBI-SS, high scores in the subscale of EX and CY indicate burnout, whereas low scores in AE indicate burnout.

SECONDARY OUTCOMES:
Jefferson Scale of Empathy-Health Profession Student version (JSE-HPS) | Baseline
  The JSE-HPS was developed with the preliminary psychometric data published in 2001 and is copyrighted by Thomas Jefferson University. The Jefferson Scale of Physician Empathy (JSPE) was originally developed to allow the measurement of empathy in physician cohorts (Hojat et al., 2001). However, given the importance of empathy as an undergraduate student trait, a number of research teams have adapted the JSPE for use with students from healthcare professions other than medicine (Fields et al., 2011; Fjortoft et al., 2011). The JSE-HPS consists of 20 items, which are responded on a seven-point Likert scale with 1 being strongly disagree and 7 being strongly agree for positively responded items and 1 being strongly agree and 7 being strongly disagree otherwise
Emotion Regulation Questionnaire (ERQ) | Baseline
  Emotion Regulation Questionnaire (ERQ) (Gross & John, 2003). This questionnaire is a 10-item self-report measure of two emotion regulation strategies: emotional suppression (ES; 4 items) and cognitive reappraisal (CR; 6 items). The participants responded on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). The total score ranged from 10 to 70 and the mean score was utilized, with a higher score presenting a higher level of emotion regulation strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Dakhlyia, Egypt

IPD SHARING:
Plan to Share IPD: No